CLINICAL TRIAL: NCT06397248
Title: DeVEnIR: Defining Vulvovaginal Candidiasis - Elements of Infection and Remedy
Acronym: DeVEnIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: KU Leuven (Other); Leibniz Institute for Natural Product Research and Infection Biology Hans Knöll Institute (Other); Universiteit Antwerpen (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 003471; S006424N (Other Grant/Funding Number: Research Foundation Flanders); 5863 (Other: Project ID - Ethical Committee UZA)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Microbiome; Innate immunity; Mycology; Infectious diseases
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * Vaginal swabs with human and microbial DNA
  * Anal swabs with human and microbial DNA
  * Buccal swabs with human and microbial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy women: Healthy volunteers that do not have vaginal complaints or symptoms, and did not have any in the past 12 months.
  Interventions: Other: No intervention
- Women with an acute episode of vulvovaginal candidiasis: Women that have sporadic/acute vulvovaginal Candida infection. It's the first time or the first time in a longer period (1-2 years) that these women have an infection.
  Interventions: Other: No intervention
- Women that suffer from recurrent episodes of vulvovaginal candidiasis: These women encounter such infections at least 3 times a year. These women are targeted both during an infection and in between infections.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Female-specific health conditions are underrepresented in research. The taboo felt by women to talk about intimate wellbeing is fed by this gender gap in scientific knowledge. This project aims to meet these needs by studying one of the most prevalent female-specific infections, vulvovaginal candidiasis (VVC), and paving the way towards its efficient diagnosis and treatment. About 70% of women worldwide suffer from vaginal candidiasis at least once in their life. An episode of this fungal infection is accompanied by a burning sensation, pain, and reduced mental well-being. Some women (about 5%) encounter such infections at least four times a year, referring to recurrent(R) VVC. The design of efficient diagnostic and therapeutic strategies for (R)VVC is hindered by a knowledge gap surrounding vaginal health. To meet the absolute need for more information, this project will characterize the role of the microbiome, metabolome, immune system, and pathogen characteristics in (R)VVC. To this end, a large sampling platform of women with/without VVC will be established in this project. The researchers will identify the most important and clinically relevant microorganisms, metabolites, and immune factors in VVC pathogenesis. VVC models will be developed and optimized, which will be used to validate the causality of the correlations identified in the cohort. Identified correlations will be proposed as biomarkers, and microbes, metabolites, and combinations, which effectively lower the pathogenicity of Candida species, will be further investigated for therapeutic potential. State-of-the-art tools and know-how of the researchers will allow the unraveling of the involved molecular pathways and elucidate how these can be exploited to optimize therapeutic efficacy. Finally, the knowledge gathered in this project will be used to improve the literacy of women on VVC using platforms established by the researchers as well as novel tools to be developed in this project.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: 18-50
* Premenopausal

Exclusion Criteria:

* Pregnancy
* Self-reported vaginal complaints (e.g. redness, itching, pain, burning sensation, abnormal vaginal discharge) in the past 12 months (only for healthy group)
* Use of antibiotics/antifungals in the month prior to sample collection (only for healthy group)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with an active Candida infection will be recruited during consultations with the responsible physicians: Prof. Gilbert Donders and Prof. Veronique Verhoeven. This subgroup will include both acute vulvovaginal candidiasis patients (episodic VVC; n=100) and recurrent VVC patients (episodic RVVC; n=100). The active Candida infection of these patients will be confirmed through clinical evaluation. Furthermore, the responsible physicians will also recruit patients who have had at least three Candida infections in the past 12 months or have already been diagnosed with RVVC. This subgroup (non-episodic RVVC; n=100) does not have an active Candida infection at the time of sample collection. Additionally, a subgroup of healthy volunteers (n=200) will be recruited through various channels. These channels will also be used to reach VVC and RVVC patients and then refer them to Prof. Donders' team.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Determining the vaginal microbial community composition of both women who suffer from (recurrent) vulvovaginal candidiasis and healthy women using Illumina MiSeq. | up to 4 years
  After metagenomic shotgun and amplicon sequencing with the Illumina MiSeq, bio-informatic tools will be used to analyze taxonomic and functional data. The researchers will specifically screen for Candida species (the main causative agent of vulvovaginal candidiasis) and other pathogenic taxa that can be associated with specific environmental conditions and lifestyle factors. Additionally, the researchers will also pay attention to health-promoting microorganisms (such as lactic acid bacteria and Saccharomyces species) that are present in the study cohort.
Determining the vaginal metabolic profile of both women who suffer from (recurrent) vulvovaginal candidiasis and healthy women using untargeted metabolomics analysis. | up to 4 years
  Swabs taken by the study cohort will be subjected to high throughput metabolomic analysis, including ultra-high performance liquid chromatography coupled with high-resolution mass spectrometry. The researchers will specifically focus on the differences in the metabolic profile of women with vulvovaginal candidiasis and healthy women. Additionally, the researchers will also pay attention to correlating these metabolic profiles with specific environmental conditions and lifestyle factors.
Determining the vaginal immunological profile of both women who suffer from (recurrent) vulvovaginal candidiasis and healthy women using multiplex ELISA assays. | up to 4 years
  Swabs taken by the study cohort will be subjected to multiplex ELISA assays. More specifically, the researchers will measure the concentration of proinflammatory cytokines known to play a role during vulvovaginal candidiasis (IL-8, IL-1a, IL-1b, IL-6, IFNa, IFNb) and compare this with data from healthy women. Additionally, the researchers will also pay attention to correlating the concentrations of proinflammatory cytokines with specific environmental conditions and lifestyle factors.
Characterizing the pathogenicity of Candida species isolated from women with vulvovaginal candidiasis using semi-high-throughput assays | up to 4 years
  Candida species isolated from the vagina of women with vulvovaginal candidiasis will be characterized for their pathogenicity. This will involve utilizing spectrophotometry, flow cytometry, and semi-automated image analysis to evaluate aspects such as growth, adhesion to epithelial cells (VK2/E6E7), and filamentation. Additionally, their capacity to cause damage will be assessed by measuring the percentage of lactate dehydrogenase released from epithelial cells through a cytotoxicity assay. Furthermore, the invasion potential of highly damaging strains will be quantified and analyzed in relation to the infection status of the women from whom the isolates were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Prof., Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - Femicare vzw, Tienen, Vlaams-Brabant
  - University of Antwerp, Antwerp

IPD SHARING:
Plan to Share IPD: Yes
The metadata of participants in the study will be made available in a restricted access repository.
  * For samples and data sharing, the researchers will work with the legal department to establish Material/Data Transfer Agreements.
  * Sequencing data are available at the European Nucleotide Archive.
  * Physical samples are their origin will be stored at the decentral hub of the Antwerp biobank.
  * Concerning non-identifiable sample meta-data that the researchers will use in analysis and will later be published will be put available with access control via the European Genome-Phenome Archive (EGA), where data can be accessed as described upon agreeing to the harmonized Data Access Agreement (developed by the European Union standards for in silico models for personalized medicine EU-STANDS4PM, https://doi.org/10.6084/m9.figshare.23904300).
Supporting Information: Study Protocol, ICF
Time Frame: Following publication, the results associated with each study will also be deposited in the Dryad repository, where they will be preserved indefinitely. Sequences will be stored to ENA (public databases) and NCBI. All samples will be registered in the Biobank using the SLIMS system. A batch of the strains will be supplied to Sciensano to be stored in the BCCM collection.
Access Criteria: A guide to data access on the EGA is available at https://ega-archive.org/access/data-access, and a data access request will be processed within 2-3 months, pending evaluation by the data access committee (existing of lab members involved in the study), and processing by the EGA.